CLINICAL TRIAL: NCT04852419
Title: A PHASE 1B STUDY TO ASSESS THE SAFETY AND TOLERABILITY OF ZN-C5 IN CHINESE SUBJECTS WITH ADVANCED BREAST CANCER
Brief Title: A PHASE 1B STUDY OF ZN-C5 IN CHINESE SUBJECTS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zentera Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: c5ZTCN100
Record Dates: First submitted 2021-04-11; First posted 2021-04-21 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Breast Neoplasms
Keywords: ER Positive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ZN-c5 50mg QD dose cohort (Experimental): Phase 1b trial of monotherapy cohort with ZN-c5 as single agent will be evaluated with ZN-c5 50 mg administered orally, once daily. Safety lead in phase will be applied.
  Interventions: Drug: ZN-c5
- Zn-c5 150mg QD dose cohort (Experimental): Once safety and tolerability are established in ZN-c5 150 mg Dose QD in Chinese population, then it is possible to initiate the second monotherapy cohort with 150 mg QD or alternative dose well established in oversea population for preliminary efficacy and safety.
  Interventions: Drug: ZN-c5

INTERVENTIONS:
Drug: ZN-c5 — ZN-c5

SUMMARY:
The aim of this phase 1b study in Chinese patients with ER+/Her2- advanced breast cancer is to evaluate the safety and tolerability of ZN-c5 at dose of 50 mg and 150 mg QD well tolerance established in the previous oversea study in non-Chinese patients.

DETAILED DESCRIPTION:
Hormone receptor-positive, HER2-negative breast cancer is the most common subset of breast cancer. The estrogen receptor (ER) in these patients is a key driver of disease progression, and the primary reason for relapse in these patients is that endocrine therapies are only partially effective, typically causing cell cycle arrest rather than cell death. As a result, secondary resistance to endocrine therapy is a major clinical challenge. ZN-c5 is a novel and potent ZN-c5 is a novel and potent selective estrogen receptor degrader with oral bioavailability and strong activity in estrogen-dependent and tamoxifen-resistant tumor models.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years
* Menopausal Status [Female subjects]
* Histologically or cytologically confirmed diagnosis of advanced adenocarcinoma of the breast, not amenable to any potential curative intervention
* Estrogen Receptor (ER) positive disease
* Human Epidermal Growth Factor Receptor 2 (HER2) negative disease
* Refractory to or intolerant of established therapy(ies) known to provide clinical benefit for their malignancy
* Prior Hormonal Therapy:
* Documented prior response to endocrine therapy for advanced or metastatic disease (SD, PR, or CR) lasting > 6 months24 weeks or disease recurrence after at least 24 months of adjuvant endocrine treatment.
* Prior Chemotherapy: Up to 2 prior lines of chemotherapy for the treatment of advanced breast cancer
* Prior treatment with a CDK4/6 inhibitor is allowed
* Evaluable or measurable disease per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1
* All acute toxic effects of any prior anti-tumor therapy resolved to Grade ≤ 1 or baseline (with the exception of alopecia [any grade permitted])
* Adequate organ function
* [Premenopausal and perimenopausal female subjects]: Negative serum pregnancy test
* Male and female subjects of childbearing potential or partners of subjects who engage in intercourse must agree to use protocol specified method(s) of contraception.

Exclusion Criteria:

* Any of the following within the specified window prior to the first dose of study drug
* Prior hematopoietic stem cell or bone marrow transplantation
* Prior radiotherapy to > 25% of bone marrow
* Brain metastases that require immediate treatment or are clinically or radiologically unstable (i.e., have been stable for < 1 month). If receiving steroids, subjects must be receiving a stable to decreasing corticosteroid dose during at least 1 week before enrollment.
* Leptomeningeal disease that requires or is anticipated to require immediate treatment.
* Presence of life-threatening metastatic visceral disease or symptomatic pulmonary lymphangitic spread
* Other known active cancer(s) likely to require treatment in the next year that would impact the assessment of any study endpoints
* [Female subjects]: Pregnant or breast-feeding
* Unexplained symptomatic endometrial disorders (including, but not limited to endometrial hyperplasia, dysfunctional uterine bleeding, or cysts)
* Impairment of gastrointestinal (GI) absorption for oral medications
* Nausea, vomiting, or diarrhea > Grade 1
* Myocardial infarction, symptomatic congestive heart failure (NYHA > Class II), unstable angina, or serious uncontrolled cardiac arrhythmia within the last 6 months
* QTc interval > 480 msec (based on the mean value of the triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or history of Torsade de Pointes
* Concurrent use of food or drugs known to be moderate or strong CYP3A or CYP2C9 inducers and moderate or strong CYP3A4 or CYP2C9 inhibitors.
* Positive serum virological tests (HBsAg, HCV-AB, HIV-AB, TP-AB) at screening stage will be excluded.
* Any clinically significant disorder, condition, or disease that, in the opinion of the Investigator or Medical Monitor would pose a risk to subject safety or interfere with the study evaluations, procedures, or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Observed Dose Limited Toxicities (DLTs) in safety lead in phase | At the end of Cycle 1 (each cycle is 28 days)
  Safety lead in phase at dose of 50 mg QD: Determine a tolerated dose for ZN-c5 in monotherapy
Incidence of treatment-emergent adverse events | until 30 days after the last dose of study drug
  Investigate the safety and tolerability of dose of 50 mg QD of ZN-c5
Incidence of treatment-emergent adverse events | until 30 days after the last dose of study drug
  Investigate the safety and tolerability of dose of 150 mg QD of ZN-c5

SECONDARY OUTCOMES:
CBR (CR [+ PR] + SD ≥ 24 weeks). | 2 year
  Investigate the preliminary antitumor activity (clinical benefit rate [CBR]) for ZN-c5 as a monotherapy using Response Evaluation Criteria in Solid Tumors (RECIST v.1.1) as assessed by investigators.
bjective Response Rate (ORR) | 2 year
  Assess preliminary antitumor activity of ZN-c5 alone by Objective Response Rate （ORR) using Response Evaluation Criteria in Solid Tumors (RECIST v.1.1) as assessed by investigators.
Duration of Response (DOR) | 2 year
  Assess preliminary antitumor activity of ZN-c5 alone by Duration of Response (DOR) using Response Evaluation Criteria in Solid Tumors (RECIST v.1.1) as assessed by investigators.
Progression-Free Survival (PFS) | 2 year
  Assess preliminary antitumor activity of ZN-c5 alone by Progression-Free Survival (PFS) using Response Evaluation Criteria in Solid Tumors (RECIST v.1.1) as assessed by investigators.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided